CLINICAL TRIAL: NCT00690794
Title: An Evaluation of the Ocular Surface Health in Subjects Using TRAVATAN Z® Ophthalmic Solution Versus XALATAN® Ophthalmic Solution
Brief Title: Travatan Z in Ocular Surface Health in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-08-03
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost (Experimental): One drop self-administered in the study eye(s) once daily for 90 days
  Interventions: Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®)
- Latanoprost (Active Comparator): One drop self-administered in the study eye(s) once daily for 90 days
  Interventions: Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®)

INTERVENTIONS:
Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 90 days. Referred to as travoprost.
  Other Names: TRAVATAN Z®
  Arms: Travoprost
Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 90 days. Referred to as latanprost.
  Other Names: XALATAN®
  Arms: Latanoprost

SUMMARY:
The purpose of the study is to compare two ophthalmic solutions in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Ocular Surface Disease Index (OSDI) score and corneal fluorescein staining score as specified in protocol.
* Diagnosis of open-angle glaucoma or ocular hypertension in at least one eye.
* Intraocular pressure (IOP) controlled with latanoprost 0.005% (XALATAN®) for at least one continuous month prior to Visit 1.
* Willing and able to discontinue use of any topical ocular medication other than the study medication for the duration of the study, including artificial tears.
* Best corrected visual acuity of -0.6 logarithm of the Minimum Angle of Resolution (logMAR) or better in each eye.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any medical condition (systemic or ophthalmic) that may preclude safe administration of the test article.
* Use of contact lenses within 30 days of Visit 1.
* Use of contact lenses during the study.
* Participation in an investigational drug or device study within 30 days of entering this study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 726 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 70 US study centers. Eligible patients having a diagnosis of open-angle glaucoma or ocular hypertension and on XALATAN® monotherapy for at least one month immediately prior to Visit 1 were enrolled.
Pre-assignment Details: 726 patients were enrolled in the study and evaluated for safety. Baseline characteristics are presented for all patients who received test article and had at least one on-therapy study visit (intent-to-treat): 678.
Period: Overall Study
Arm/Group | Travoprost | Latanoprost
Started | 363 | 363
Completed | 342 | 328
Not Completed | 21 | 35
Not completed — Adverse Event | 12 | 10
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 0 | 9
Not completed — Protocol Violation | 6 | 7
Not completed — Noncompliance | 1 | 2
Not completed — Other not specified | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost | Latanoprost | Total
Number analyzed (Participants) | 343 | 335 | 678
Age Continuous [Mean (Standard Deviation); unit: years] | 67.1 (11.0) | 67.8 (10.8) | 67.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 230 | 441
  Male | 132 | 105 | 237

OUTCOME MEASURES:

1. Primary Outcome: Mean Change at Day 90 From Baseline (Day 0) in Ocular Surface Disease Index (OSDI) Score
Description: The OSDI is a 12-question validated questionnaire (resultant overall 0-100 point score) used to measure ocular symptoms, visual function and environmental factors that may affect a patient's vision, where 0 = normal and 100 = severe. The OSDI questionnaire was administered at both visits and completed by the patient with no assistance from the office staff, physician, or anyone else. The baseline OSDI score was subtracted from the 90-day OSDI score and reported as change. A negative number represents a perceived improvement in ocular health.
Time Frame: Baseline, Day 90
Population: Intent-to-treat. All patients who received test article and had at least one on-therapy study visit were evaluable for the intent-to-treat analysis. An Observed Case analysis (OC) was performed for the ITT population.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 339 | 328
Units on a scale | -11.3 (0.9) | -11.4 (1.0)

2. Secondary Outcome: Percentage of Patients With Corneal Fluorescein Staining Score = 0
Description: The corneal surface was assessed by the investigator and graded on a scale of 0-3, where 0 = Absent (no staining present) and 3 = Severe (>50% coverage). Percentage of patients with score = 0 at 90 days was calculated by dividing the number of patients with score = 0 by the total number of patients analyzed.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 342 | 330
percentage of patients | 37.1 | 40.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 03 July 2008 to 26 May 2009.
Description: This reporting group includes all patients who received the test article.
Arm/Group | Travoprost | Latanoprost
Serious Adverse Events (participants affected / at risk) | 5/363 | 7/363
Other Adverse Events (participants affected / at risk) | 0/363 | 0/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Travoprost (N=363) | Latanoprost (N=363)
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Brachycardia (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The subjective nature of the OSDI may not be sensitive enough to detect the effects of preservatives on the corneal surface. The measurement and quantification of OSD remains a considerable clinical challenge. (Pflugfelder and Baudoin, 2011)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.